CLINICAL TRIAL: NCT02858284
Title: A Multi-Center, Randomized, Double-Masked, 8-week Pilot Study Evaluating the Safety and Efficacy of the TUG (Therapeutic Ultrasound for Glaucoma) Compared to Sham in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Evaluation of Safety and Efficacy of TUG (Therapeutic Ultrasound for Glaucoma) in the Treatment of Primary Open Angle Glaucoma or Ocular Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor request
Sponsor: EyeSonix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUG-US-001
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2019-02

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TUG Device (Experimental): 1 time external application - device powered on
  Interventions: Device: TUG
- Sham (Sham Comparator): 1 time external application - device powered off
  Interventions: Device: Sham

INTERVENTIONS:
Device: TUG — Therapeutic Ultrasound for Glaucoma
  Arms: TUG Device
Device: Sham
  Arms: Sham

SUMMARY:
The purpose of this study is to evaluate whether the TUG device is safe and effective in patients with primary open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of primary open angle glaucoma or ocular hypertension in both eyes
* Be willing to discontinue disallowed products and/or medications during the period indicated prior to participation or throughout the study
* Be willing to provide written informed consent
* Be willing and able to follow instructions
* A negative urine pregnancy test and agree to an acceptable form of contraception for the duration of the study (if female of childbearing potential)

Exclusion Criteria:

* Any form of glaucoma other than primary open angle glaucoma or ocular hypertension in either eye
* Prior or anticipated concurrent use of an investigational drug or device
* Be currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive pregnancy test
* Have a condition (ocular or systemic) or a situation which, in the Investigator's opinion, may put the subject at increased risk, may confound study data, or may interfere significantly with the subject's study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Change in mean IOP | through subject study completion; average 2 months
Change in mean diurnal IOP | Week 4 (Visit 5) and Week 8 (Visit 7)
Change in IOP from baseline | through subject study completion; average 2 months